CLINICAL TRIAL: NCT02656342
Title: Translational Approach to the Understanding and Treatment of Obsessive-Compulsive Disorder (OCD). Can D-Cycloserine Enhance and Stabilize the Treatment-response in Relapsed and Non-responding OCD-patients? A Randomized, Double-blind, Placebo-controlled National Study
Brief Title: Translational Approach to the Understanding and Treatment of Obsessive-Compulsive Disorder (OCD). Can D-Cycloserine Enhance and Stabilize the Treatment-response in Relapsed and Non-responding OCD-patients?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Helse Vest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-002574-49
Record Dates: First submitted 2015-11-30; First posted 2016-01-14 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 250 mg DCS (Experimental): 64 patients receive 250 mg D-Cycloserine two consecutive days in combination with therapist assisted concentrated exposure therapy (cET)
  Interventions: Drug: D-Cycloserine
- 100 mg D-Cycloserine (Experimental): 64 patients receive 100 mg D-Cycloserine two consecutive days in combination with therapist assisted concentrated exposure therapy (cET)
  Interventions: Drug: D-Cycloserine
- Placebo (Active Comparator): 32 patients receive placebo two consecutive days in combination with therapist assisted concentrated exposure therapy (cET)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine — Predicted to enhance stabilization of the effects of concentrated exposure treatment
  Other Names: DCS; Cycloserine
  Arms: 100 mg D-Cycloserine; 250 mg DCS
Drug: Placebo — Predicted to have no enhancing effect
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
In this randomized controlled trial (RCT) the investigators experimentally test if patients with Obsessive-Compulsive Disorder (OCD) who have received treatment with exposure and response prevention (ERP), but either relapsed or not responded, profit from the combination of concentrated exposure based treatment (cET) and the NMDA-agonist (N-methyl-d-aspartate) d-cycloserine (DCS), targeting fear relevant areas in amygdala and pre-frontal cortex.

The project expects to demonstrate a significant improvement in all groups, and anticipate that a higher proportion of the patients who receive DCS will show a better long-term gain from the treatment, as compared to the placebo group at follow-up (3 mon, 12 mon, and 5 years after treatment). In addition, the project will highlight changes in depression, sleep, global functioning, quality of life, work and social status. Changes in medication and use of health care will be included and related to the main objective of the study.

DETAILED DESCRIPTION:
A total of 160 relapsed and non-responding OCD-patients, treated with exposure and response prevention (ERP) in the specialist Health care in Norway, are planned to participate in the study: "Translation approach to the understanding and treatment of Obsessive-Compulsive Disorder (OCD). Can D-cycloserine (DCS) enhance and stabilize the treatment-response in relapsed and non-responding OCD-patients? A randomized, double-blind, placebo-controlled national study." Estimated start of inclusion is November 2015 and the inclusion period lasts for maximum 2 years. All participants are referred to the specialist health care and are pre-screen by the local OCD-team. Before inclusion, the patients will fill in a number of questionnaires on-line and all patients who meet the inclusion criteria will be invited to participate. Before the patient signs the informed consent form the patients will receive written and oral information about the study as well as watch a video describing the trial and what participation will imply. Before the 4-day concentrated exposure based treatment (cET) starts, the patients will undergo a clinical assessment interview by the local OCD-team, and will watch another video describing the trial in detail. They will also be assessed by SCID-I (Structured Clinical Interview) for DSM 5 as well as Y-BOCS (Yale-Brown Obsessive Compulsive Scale) interview by independent and specially trained psychologists. The cET is delivered in an "individual group format" which implies that the patient: therapist-ratio is 1:1, and that the treatment is delivered in groups of minimum 3 and maximum 6 patients. All groups are led by a specially trained cET therapist, and the local therapists are experienced OCD-therapists who are familiar with the cET format. Day 1 of the treatment (3 h) consists of psychoeducation and planning of exposure tasks. Day 2 and day 3 (both 8 h + contact in the evening) consist of individually tailored and therapist assisted exposure with a number of relevant triggers in a diversity of settings. All exposures are based on the LEaning in Technique (LET), where the patients are trained to recognize when the urge to ritualize starts, and to actively approach the trigger by "leaning into the anxiety". The exposures are also designed to optimize learned inhibition. In addition to individual exposure training, the group meets three times throughout the day. Day 2 and Day 3 the patient will take study medication before the exposures start. The study medication is D-Cycloserine (DCS) 250 mg, DCS 100 mg or placebo. In the afternoon Day 3, the patients' relatives/ friends are invited to a 2 h lecture/ psychoeducation on OCD and the current treatment. Day 4 the focus is on "lessons learnt" as well as on planning / specifying exposure tasks for the coming three weeks. Before and during the cET the patient will record data electronically via CheckWare (an electronic case report form database). The patient will continue registration of obsessions and compulsions through 3 weeks post cET. One week after cET a post-assessment with Y-BOCS will be performed by the independent assessor. After 3 months, the patient is invited to an individual visit at the clinic. 1 year and 5 years post treatment, the assessment team will perform follow-up telephone interviews.

Measures of anxiety, depression, global functioning, severity of the disorder, self-reported OCD-symptoms, sleep, quality of life, changes in work and social status as well as changes in medication and use of health care will be included and employed as secondary outcomes.

A total of 14 expert therapists have been trained to deliver cET to OCD-patients all over Norway. Patients, therapists and assessors are all blinded to the randomization. Interventions are recorded and rated for compliance and competence . All SCID-I and Y-BOCS assessments are recorded and standard procedures for rescoring are followed. All assessors are independent and specially trained.

A Scientific Advisory Board is established, also including representatives from the Norwegian OCD-association. The formal project partners are Haukeland University Hospital; Oslo University Hospital; St Olavs Hospital; Soerlandet Hospital and Moere and Romsdal Hospital.

ELIGIBILITY:
All 15 OCD-teams in Norway refer patients to the study, thus providing nationwide coverage of relapsed or non-responsive OCD patients.

Through the Norwegian National OCD-implementation project all OCD-patients in Norway are ensured access to evidence based treatment. Standardized procedures for collection and storage of data (quality databases) are also established. These data will serve as reference data for standard treatment response, as well as provide detailed information regarding the first treatment-course for the relapsed OCD-patients.

The inclusion procedure implies that all relevant patients in Norway in the given time period will be offered participation. If this population turns out to be fewer than 160 patients during the study period, the inclusion period might be extended six months. If less than 160 patients are included at that point, analyses will be performed on the number of patients included by the end of the study period.

Inclusion Criteria:

* Outpatients
* ≥ 18 years
* Fulfilling diagnostic criteria of OCD according to the DSM-5
* Previously have received ERP-treatment delivered by trained therapist and either have responded and relapsed, or not responded to the treatment.
* Response is defined by ≥35% reduction with a post-treatment Y-BOCS score of ≤15, followed by a relapse as defined by > 35% increase in Y-BOCS score from post-treatment, a Y-BOCS score of 16 or more, and a Clinical Global Impression-Improvement Scale (CGI-I) score of 6 ("much worse") or higher.
* Non-responders are defined as those with a reduction in Y-BOCS scores from pre- to post-of less than 35%, and with a Y-BOCS score of ≥16 after treatment. In order to be classified as non-responder as opposed to "drop-out" the patient has to previously have received a minimum of 6 sessions.
* There must be a minimum of 4 weeks since treatment ended.
* Fluent in Norwegian
* Signed informed consent

Exclusion Criteria related to the ERP:

* OCD symptoms primarily associated with hoarding
* Ongoing substance abuse/dependence
* Bipolar disorder or psychosis
* Ongoing suicidal ideation
* Mental Retardation, based on previous medical history
* If using antidepressants:
* Not on stable dosage 12 weeks before the intervention
* Unwilling to remain on stable dosage during the four intervention days
* Unwilling to refrain from anxiolytics (e.g. benzodiazepines) and alcohol during the two days of exposure.
* Living > 1 hour drive by car/ train from the treatment location.

Exclusion Criteria related to the DCS:

* Pregnancy or breast feeding (the participants are informed that they will have to use contraception the two days when the DCS/placebo is administered. Females will be asked if they are pregnant, and in case of doubt a pregnancy test is provided)
* Renal impairment
* Hypersensitivity to D-Cycloserine
* Porphyria
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Changes in Y-BOCS | 3 and 12 months, 5 years
  Response is a ≥35% reduction of the individual patient's pre-treatment YBOCS score. A patient is remitted if the response criterion is fulfilled and the post-treatment Y-BOCS score is ≤12
Changes in diagnostic status | 3 and 12 months, 5 years
  Changes in Diagnostic status (DSM-5) assessed by SCID-I for DSM-5 at above specified points.
Changes in Y-BOCS evaluated by Jacobson and Truax, Reliable Change Index (RCI) | 3 and 12 months, 5 years
  The criteria of Jacobson and Truax: A.Change from pre- to post-assessment is statistically reliable at the 5%-level. (RCI). B. The patient's post-treatment score is within the distribution of the normal population defined as M+2Standard Deviation (SD), or outside the distribution of the patient population defined as M-2SD. Non-responder is not fulfilling the RCI. Partial responder fulfills the RCI but not the cut-off score Full responder fulfils the RCI and the cut-off score.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Kvale, Principal Investigator — Haukeland University Hospital; Bjarne Hansen, Principal Investigator — Haukeland University Hospital; Michelle Craske, PhD, Study Chair — Haukeland University Hospital; Jonathan Abramowitz, PhD, Study Chair — Haukeland University Hospital; Hime A Joeseph, PhD, Study Chair — Haukeland University Hospital; Martin D Franklin, PhD, Study Chair — Haukeland University Hospital; Michael Davis, PhD, Study Chair — Haukeland University Hospital; Lars-Göran Öst, PhD, Study Chair — Haukeland University Hospital; Odile van den Heuvel, PhD, Study Chair — Haukeland University Hospital
Locations (14):
- Norway (14):
  - Haukeland University Hospital, Bergen
  - Innlandet Hospital, Brumunddal
  - Forde Hospital, Førde
  - Sørlandet Hospital, Kristiansand
  - Nord Trøndelag Hospital, Levanger
  - Akershus University Hospital, Lorenskog
  - More and Romsdal Hospital, Molde
  - Østfold Hospital, Moss
  - Oslo University Hospital, Oslo
  - Vestre Viken, Sandvika
  - Stavanger University Hospital, Stavanger
  - Tromso University Hospital, Tromsø
  - St. Olavs Hospital, Trondheim
  - Sykehuset i Vestfold, Tønsberg

REFERENCES:
- [Derived] Tjelle K, Hansen B, Solem S, Wheaton MG, Kvale G, Hagen K. Concentrated ERP for Patients With Difficult-to-Treat OCD: Insight as a Predictor of Acute and Long-Term Outcomes. Depress Anxiety. 2025 Dec 11;2025:8960147. doi: 10.1155/da/8960147. eCollection 2025. PMID 41425659
- [Derived] Berg H, Tjelle K, Hansen B, Solem S, Bjorgvinsson T, Kvale G, Hagen K. Treatment expectancy and credibility as predictors of concentrated exposure treatment outcomes in patients with difficult-to-treat obsessive-compulsive disorder. BMC Psychiatry. 2025 Mar 25;25(1):275. doi: 10.1186/s12888-025-06737-z. PMID 40133857
- [Derived] Tjelle K, Opstad HB, Solem S, Kvale G, Wheaton MG, Bjorgvinsson T, Hansen B, Hagen K. Patient adherence as a predictor of acute and long-term outcomes in concentrated exposure treatment for difficult-to-treat obsessive-compulsive disorder. BMC Psychiatry. 2024 Apr 30;24(1):327. doi: 10.1186/s12888-024-05780-6. PMID 38689256
- [Derived] Kvale G, Hansen B, Hagen K, Abramowitz JS, Bortveit T, Craske MG, Franklin ME, Haseth S, Himle JA, Hystad S, Kristensen UB, Launes G, Lund A, Solem S, Ost LG. Effect of D-Cycloserine on the Effect of Concentrated Exposure and Response Prevention in Difficult-to-Treat Obsessive-Compulsive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2013249. doi: 10.1001/jamanetworkopen.2020.13249. PMID 32789516
- See also: Homepage for the OCD-team i nBergen and the national OCD-study — http://www.helse-bergen.no/ocd